CLINICAL TRIAL: NCT01694602
Title: Non-Invasive Assessment of Skeletal Muscle Loss in Cancer Patients - Phase 2
Brief Title: Non-Invasive Assessment of Skeletal Muscle Loss in Cancer Patients - Phase II
Acronym: 3MH-2
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 12-064; 2R44AR054993-02 (NIH)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Cachexia
Keywords: Cachexia; Sarcopenia; De Novo; Deuterated
MeSH Terms: conditions — Cachexia; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Spot urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly Diagnosed NSCLC patients: In this study, newly diagnosed NSCLC patients who are not candidates for curative resection, will receive a (non-radioactive) oral dose of deuterated 3-methylhistidine (D-3MH).
  Interventions: Biological: (non-radioactive) Oral deuterated 3-methylhistidine (D-3MH)

INTERVENTIONS:
Biological: (non-radioactive) Oral deuterated 3-methylhistidine (D-3MH) — Oral dose of 9.0 mg (50 μmol) TAU-METHYL-L-HISTIDINE (METHYL-D3), Cambridge Isotope Laboratory, Cambridge, Massachusetts.

SUMMARY:
The overall aim of this research is to develop a non-invasive approach to evaluate the production of 3-methylhistidine (3MH)in cancer patients, as a potential means of determining which patients are at high risk for future development of cancer induced skeletal muscle atrophy.

Rationale: The approach is based on the hypothesis that after an oral dose of deuterated 3-methylhistidine (D-3MH), the slope of the terminal portion of the decay curve (> 12 hours post-dosing) for the tracer/tracee (D-3MH/3MH) in the free 3MH pool is proportional to the rate constant for myofibrillar protein degradation and can be determined from spot urine samples.

DETAILED DESCRIPTION:
The long-term objective of this research is to develop a non-invasive approach for assessment of de novo 3MH production in cancer patients early in the course of the disease as a way of assessing which patients are at high risk for future development of skeletal muscle atrophy. The approach is based on: 1) the known increase in de novo production of 3-methylhistidine (3MH) from muscle protein breakdown in said patients as a consequence of their unique disease-host interactions, and 2) earlier demonstration that de novo 3MH production can be measured in vivo using isotope dilution.

During this Phase-II project, we propose to conduct a statistically powerful prospective investigation to demonstrate that measurement of the slope of the terminal decay curve (rate constant) with our approach in newly diagnosed cancer patients predicts future development of muscle wasting. We expect the outcome of the combined Phase-I and Phase-II research to lead to the early identification of elevated muscle catabolism in at-risk patients so that medical intervention can prevent future muscle atrophy.

ELIGIBILITY:
Inclusion Criteria:

* (1) histological or cytological evidence of NSCLC without curative options;
* (2) over 18 years of age;
* (3) patient reported weight loss of ≤5% of usual body weight in the last 6 months;
* (4) life expectancy of greater than 6 months based on the judgement of treating physician;
* (5) serum creatinine ≤1.5 times the upper limit of normal; and
* (6) willing and able to give informed consent.

Exclusion Criteria:

* 1) malabsorption, intractable vomiting or gastrointestinal obstruction
* 2) congestive heart failure
* 3) edema or ascites
* 4) liver function test results that will preclude administration of prescribed therapy
* 5) pregnant, nursing, or, if of child-bearing age, unwilling to use contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will conduct a longitudinal study (repeated measures design) in 30 newly diagnosed nonsmall cell lung cancer (NSCLC) patients who are not candidates for curative resection.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determination of myofibrillar protein degradation rate constant and slope of terminal decay curve. | Spot urine (multiple) collections between 12 to 17 hours of D-3MH ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: William J Durham, PhD, Principal Investigator — The University of Texas Medical Branch (UTMB Health), Galveston, Texas.
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States